CLINICAL TRIAL: NCT02599493
Title: EVRIOS : Comparative Evaluation of Low Versus High Doses of Rifampicin in the Treatment of Staphylococcal Bone and Joint Infections
Brief Title: EVRIOS : Comparative Evaluation of Low Versus High Doses of Rifampicin
Acronym: EVRIOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35RC14_9741_EVRIOS; 2015-001519-11 (EudraCT Number); 150790A-41 (Other: ANSM); 15/18-980 (Other: CPP)
Record Dates: First submitted 2015-11-03; First posted 2015-11-06 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Osteoarticular Infection
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose (Experimental): Patients will be randomly assigned to low dosage (10 mg/kg/j) rifampicin group. Rifampicin treatment will be prescribed in association with another antibiotic chosen by investigator according to the antibiogram results. Association with fluoroquinolones is the first choice combination, if it is possible. The global antibiotic treatment duration depends on the investigator's choice.
  Interventions: Drug: Rifampicin
- High dose (Active Comparator): Patients will be randomly assigned to high dosage (20 mg/kg/j) rifampicin group. Rifampicin treatment will be prescribed in association with another antibiotic chosen by investigator according to the antibiogram results. Association with fluoroquinolones is the first choice combination, if it is possible. The global antibiotic treatment duration depends on the investigator's choice.
  Interventions: Drug: Rifampicin

INTERVENTIONS:
Drug: Rifampicin — Patients will be randomly assigned to low dosage (10 mg/kg/j) rifampicin group or high dosage (20 mg/kg/j) rifampicin group. Rifampicin treatment will be prescribed in association with another antibiotic chosen by investigator according to the antibiogram results. Association with fluoroquinolones is the first choice combination, if it is possible. The global antibiotic treatment duration depends on the investigator's choice.
  Other Names: RIMACTAN

SUMMARY:
Rifampicin is an antibiotic usually required to treat susceptible Staphylococcus spp. osteo-articular infections, most frequently in association with a fluoroquinolone when the strain is susceptible to both agents. It is the reference treatment for orthopedic infections with implanted material.

For tuberculosis treatment the dosage of 10 mg/kg/j is usually prescribed, while in the treatment of Staphylococcus spp. infections the highest dosage of 20 mg/kg/j is proposed by French experts' recommendations from 2009.

However, there is little evidence in the literature, which could set out arguments to choose the best dosage of rifampicin, which may vary from 5 to 20 mg/kg.

The issue with rifampicin is side effects, in particular with long-term treatment. Many side effects may occur in 10 to 20% of patients and sometimes leads to dosage reduction or treatment interruption.

In the literature, there is little evidence that higher rifampicin dosage is associated with higher frequency of adverse effects. Depending on the nature of the toxicity, one could say that hypersensitivity could be independent from dosage, when digestive disorders may be related. Plasmatic concentrations studies have not given strong arguments to link higher rifampicin dosages with side effects occurrence rates. After oral absorption, plasmatic peak occurs after two to five hours and varies among individuals but also in the same patient overtime. This particular pharmacokinetic profile could explain discrepancy in adverse events (AEs) frequencies.

DETAILED DESCRIPTION:
Primary objective :

To demonstrate that a daily weight-based low dose of rifampicin is non-inferior to a high dose in the treatment of susceptible Staphylococcus spp. osteo-articular infections.

Secondary objectives :

To compare, in the two treatment groups (weight-based low dose rifampicin versus weight-based high dose):

* Possible failure rates (when no bacteriological samples are available or when clinical manifestations are not straightforward),
* AEs distribution:

  * Those self-patient reported,
  * Those medical or biological reported,
* - Rifampicin dose modifications:

  * Dosage decrease,
  * Treatment interruption (temporary or definitive),
* Failure risk factors analysis,
* Health costs related to the osteo-articular infection care: number and length of hospitalizations, number of follow-up visits, nature and number of all biological samples prescribed in both groups.
* Comparison of the planned rifampicin exposure in each randomization group
* Differences in rifampicin duration (planned versus effective duration) according to allocated group,
* Rifampicin pharmacokinetics sub-study in a small sample of 60 patients,
* Rifampicin resistance bacteriological study in patients with proven failure.

Methodology :

Non-inferiority prospective, multicentre, randomized, open-label, controlled phase IV trial evaluating two different rifampicin dosages (high versus low dose) in the treatment of staphylococcal bone and joint infections.

Treatment :

Patients will be randomly assigned to low dosage (10 mg/kg/j) rifampicin group or high dosage (20 mg/kg/j) rifampicin group. Rifampicin treatment will be prescribed in association with another antibiotic chosen by investigator according to the antibiogram results. Association with fluoroquinolones is the first choice combination, if it is possible. The global antibiotic treatment duration depends on the investigator's choice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years old) who gave their signed inform consent,
* Who present an osteo-articular infection with susceptible Staphylococcus spp.,
* To whom a rifampicin based regimen is prescribed, in association with another antibiotic, for at least 14 days,
* Patients covered by Health Insurance.

Exclusion Criteria:

* Patients weighing less than 45 kg or more than 150 kg,
* Patients with active TB (whatever its localization),
* Patients needing the imperative use of a treatment presenting a contraindication for concomitant use in the SPC of Rimactan®
* Patients with a known and documented rifampicin allergy or severe rifampicin intolerance,
* Patients with galactose intolerance, total lactase deficiency or glucose or galactose malabsorption syndrome, or any other contraindication to the administration of Rimactan® listed in the SPC for Rimactan®
* Pregnant or breastfeeding woman,
* Adults legally protected (under judicial protection, guardianship or supervision), persons deprived of their liberty,
* Patients participating in another interventional clinical trial (biomedical trial or standard care clinical trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2016-01; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Proven failure | 12 months
  The rate of proven failure between the two groups, 12 months after the end of antibiotics.
  The proven failure is defined as a documented bacteriological failure, with the same Staphylococcus spp. strain isolated before the onset of antibiotics and at diagnosis of failure.

SECONDARY OUTCOMES:
Possible failure | 12 months
  Possible failure rates: defined as the lack of documented bacteriology and presence of septic clinical manifestations according to French experts recommendations.
Adverse events | 12 weeks
  Biological and clinical AEs.
Dose modification | 12 weeks
  Rifampicin dose modification: each rifampicin dosages change or interruption.
Failure risk factors | 12 months
  Failure risk factors: collected for each patient and include those already known in the literature: bacterial strains type, anatomic site of infection, presence of prosthetic material, duration of infectious signs, waiting period between first infectious signs and medical care, type of surgical intervention (with or without prosthetic material removal), type, duration and administration road of antibiotics treatment, patient's age, concomitant pathologies.
Global health costs | 12 weeks
  Global health costs: rhythm of visits defined by investigator site until the end of antibiotic treatment, all additional visit and/or exams or concomitant treatment prescriptions will be collected at each schedule visit, analysed and compared in two groups of rifampicin treatment.
Real antibiotics treatment duration | 12 weeks
  Real antibiotics treatment duration
Plasma concentration | 12 hours
  Rifampicin Pharmacokinetic: it will be studied in a sub-sample of 60 patients (30 in each group) at the onset of rifampicin-based regimen and will estimate rifampicin plasmatic concentration, self-induction mechanism and possible links with ARs or adverse occurrences.
Staphylococcus spp. resistance | 12 months
  Analysis of Staphylococcus spp. resistance: in case of proven failure, will compare strains in the same patient and resistant strains incidence into the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Cédric ARVIEUX, MD, Principal Investigator — Rennes University Hospital
Locations (16):
- France (16):
  - Angers university hospital, Angers
  - Bordeaux university hospital, Bordeaux
  - Brest university hospital, Brest
  - Caen university hospital, Caen
  - La Roche sur Yon hospital, La Roche-sur-Yon
  - Lorient hospital, Lorient
  - Clinique du Parc et Hôpital Jean Mermoz, Lyon
  - Nantes university hospital, Nantes
  - Pau hospital, Pau
  - Poitiers university hospital, Poitiers
  - Rennes university hospital, Rennes
  - Saint-Brieuc hospital, Saint-Brieuc
  - Saint-Malo hospital, St-Malo
  - Toulouse university hospital, Toulouse
  - Tours university hospital, Tours
  - Vannes hospital, Vannes